CLINICAL TRIAL: NCT04504526
Title: Value of Chemokine Receptor CXCR4-targeting Molecular Imaging for Diagnosis and Prognostic Evaluation in Lymphoproliferative Diseases
Brief Title: Value of Chemokine Receptor CXCR4 Imaging for Diagnosis and Prognostic Evaluation in Lymphoproliferative Diseases
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, Weibing Miao, PhD, Director of Nuclear Medicine Department, First Affiliated Hospital of Fujian Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FirstAHFMUCXCR4
Record Dates: First submitted 2020-08-01; First posted 2020-08-07 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-02

CONDITIONS: Lymphoma; Multiple Myeloma; Leukemia
MeSH Terms: conditions — Lymphoma; Multiple Myeloma; Leukemia | interventions — 68Ga-pentixafor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-Pentixafor, PET/CT (Experimental): PET/CT perform after injecting 68Ga-Pentixafor
  Interventions: Drug: 68Ga-Pentixafor

INTERVENTIONS:
Drug: 68Ga-Pentixafor — Intravenous injection of one dose of 74-148 MBq (2-4 mCi) 68Ga-Pentixafor. Tracer doses of 68Ga- Pentixafor will be used to image lesions by PET/CT.

SUMMARY:
Chemokine receptor CXCR4 is normally expressed on T-lymphocytes, B-lymphocytes, monocytes, macrophages, neutrophils and eosinophils as well as hematopoietic stem and progenitor cells (HSPC) in the bone marrow. 68Ga-Pentixafor PET/CT represents a promising method for the in vivo assessment of the CXCR4 expression status in cancer patients, especially in hematologic malignancies. This prospective study is going to investigate whether metabolic characterization by 68Ga-Pentixafor PET/CT may be superior for diagnosis, risk stratification, and the prognostic evaluation in lymphoproliferative diseases.

DETAILED DESCRIPTION:
Lymphoma:

The marginal zone lymphoma, plasma cell lymphoma, T-cell-lymphoma frequently do not present with an elevated FDG uptake. However, lymphoma is a frequent cancer with high CXCR4 expression. The previous studies showed 68Ga-pentixafor-PET seems to be a highly selective and specific method for the in vivo quantification of CXCR4 expression. Thus, our study is going to investigate the value of 68Ga-pentixafor-PET/CT for the diagnosis and prognostic evaluation of CXCR4 expression in lymphoma.

Multiple myeloma:

Multiple myeloma (MM) is characterized by the neoplastic proliferation of plasma cells producing a monoclonal immunoglobulin. Minimal residual disease (MRD) status is an important predictor of clinical outcome in MM. But it is difficult to assess the accurate MRD status because of the significant heterogeneity characterizing with 18F-FDG PET/CT. Studies showed Chemokine receptor CXCR4 was expressed in MM cells and CXCR4-targeting molecular imaging-68Ga-Pentixafor PET/CT could be a promising technique to evaluate the extent of MM with higher accuracy. This prospective study is going to investigate the value of 68Ga-Pentixafor PET/CT for the diagnosis and prognostic evaluation of CXCR4 expression in MM.

Leukemia： Leukemia is the second largest family of hematological malignancies after the lymphomas, and, depending on the subtype, may show a considerable overlap of histological features with the latter. The four main kinds of leukemia are, in the order of their prevalence. Imaging has traditionally played a limited role in the work-up of leukemias, with regard to detection, staging, and response assessment. 18F-FDG PET/CT is not recommended for routine evaluation of CLL, because the disease shows low uptake in the majority of cases. Although, the clinical utility of MRI lies in the detection of bone marrow abnormalities that are suspicious for leukemia in adult and pediatric patients with unclear musculoskeletal symptoms with its reduced radiation dose (in comparison with PET/CT). However, it may become more attractive with the use of newer, non-FDG PET radiotracers. High CXCR4 expression is known to be associated with poor prognosis in CLL. Recently, the feasibility of 68Ga-Pentixafor PET has also been demonstrated for CLL and AML. This prospective study is going to investigate the value of 68Ga-Pentixafor PET/CT for the diagnosis and prognostic evaluation of CXCR4 expression in leukemia.

ELIGIBILITY:
Inclusion Criteria:

* suspected or confirmed untreated Lymphoproliferative diseases patients
* 18F-FDG PET/CT within two weeks
* signed written consent.

Exclusion Criteria:

* pregnancy
* breastfeeding
* known allergy against Pentixafor

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-08-07 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
SUVmax | through study completion, an average of 3 years
  SUVmax of focal lesions are measured on 68Ga-Pentixafor PET/CT. The SUVmax of the liver, and/or mediastinal blood pool, and/or L3 vertebra are defined as the background.
The time for patient's survival | through study completion, an average of 3 years
  Investigators follow up and record the time for patient's survival. To investigate the ralationship between initial SUVmax of focal lesions and survival. Finally, the prognostic evaluation of 68Ga-Pentixafor PET/CT for lymphoproliferative diseases in comparison with 18F-FDG PET/CT.

SECONDARY OUTCOMES:
Diagnostic sensitivity and specficity in special type of lymphoma | through study completion, an average of 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Weibing Miao, M.D., Principal Investigator — First Affiliated Hospital of Fujian Medical University
Locations (1):
- Department of Nuclear Medicine, First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pan Q, Chen Z, Liu S, Zhang H, Feng J, Miao W, Li F, Cao X, Luo Y. Reduced splenic uptake of [68Ga]Ga-Pentixafor following first-line chemotherapy is associated with poor prognosis in patients with newly diagnosed multiple myeloma. EJNMMI Res. 2025 Jun 20;15(1):74. doi: 10.1186/s13550-025-01262-2. PMID 40540129
- [Derived] Chen Z, Yang A, Zhang J, Chen A, Zhang Y, Huang C, Chen S, Yao S, Miao W. CXCR4-Directed PET/CT with [68Ga]Pentixafor in Central Nervous System Lymphoma: A Comparison with [18F]FDG PET/CT. Mol Imaging Biol. 2022 Jun;24(3):416-424. doi: 10.1007/s11307-021-01664-3. Epub 2021 Oct 14. PMID 34651291